CLINICAL TRIAL: NCT00177749
Title: Open Label, Limited Access Protocol of Posaconazole in Invasive Fungal Infections Study PO2095
Brief Title: Limited Access Protocol of Posaconazole in Invasive Fungal Infections Study PO2095
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study is complete Analysis is complete
Sponsor: University of Pittsburgh (Other)
Collaborators: Schering-Plough (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB#0307071
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Fungal Infection
Keywords: invasive fungal infections
MeSH Terms: conditions — Mycoses; Invasive Fungal Infections | interventions — posaconazole

INTERVENTIONS:
Drug: Posaconazole

SUMMARY:
Therapeutic options for serious fungal infections are limited by intrinsic and acquired resistance to existing antifungal agents. For example, zygomycetes (such as Mucor spp.) are intrinsically resistant to voriconazole and caspofungin. Yet, the only available therapeutic option, amphotericin, is associated with significant renal toxicity, even in lipid formulations. Posaconazole is a new antifungal drug, not yet Food and Drug Administration (FDA) approved, but which has excellent in vitro activity against some intrinsically resistant fungi such as the zygomycetes.

The intent of this trial is to provide access to posaconazole to patients with serious fungal infections which are refractory to standard antifungal therapies or invasive fungal infections for which there are currently no effective therapies. Secondly, the drug will also be made available to patients with invasive fungal infections who:

* have experienced serious or severe toxicities while receiving standard antifungal therapies;
* have pre-existing renal dysfunction which precludes use of standard antifungal therapies; or
* are chronically immunosuppressed with a history of invasive fungal infections previously treated with posaconazole in other clinical trials, and who require oral antifungal suppressive therapy as maintenance treatment to prevent recurrence.

This is a multicenter, open-label, non-comparative experimental treatment use protocol. The experimental treatment use protocol will provide the investigational medication posaconazole where no other drug is commercially available. Posaconazole is given as an orally or enterally administered suspension. The duration of therapy is at the discretion of the investigator. Safety assessments will include an electrocardiogram [ECG] (to ensure no QTc interval prolongation) performed at baseline and serum/urine pregnancy testing performed at baseline and every three months after initiation of therapy. Plasma concentrations will be obtained if there is evidence of clinical failure. No other tests will be performed specifically for the experimental treatment use protocol.

DETAILED DESCRIPTION:
This is an open-label, multi-center limited access experimental treatment use protocol of Posaconazole in the treatment of Invasive Fungal Infections. This experimental treatment use protocol is projected to begin enrollment in September 2001.

Screening:

1. complete medical history, including a review of the subject's fungal infection and the antifungal treatment(s)
2. women of childbearing potential, will have a serum (blood) or urine pregnancy test before the experimental medication (posaconazole) is administered. This test requires a sample of blood to be drawn (10 mL or 1 tablespoon of blood or about 10 ml or 1 tablespoon of urine). The subject will not be able to participate in this experimental treatment use protocol if pregnant. In addition, while participating in this experimental treatment use protocol, women of childbearing potential, will have serum (blood) or urine pregnancy tests performed every 3 months.
3. Electrocardiogram- ECG

The total time for all these screening tests will be one hour and will be carried out in the subject's hospital room.

Experimental Procedures: the following procedures that are not part of the subject's standard medical care. This experimental treatment use protocol will be conducted worldwide. This experimental treatment use protocol is open ended so no set subject enrollment has been set by Schering Plough. It is anticipated that sites may be opened for a single patient, and we anticipate enrolling up to two patients at UPMC. All subjects enrolled in this open-label experimental treatment use protocol will receive treatment with posaconazole as outlined previously. Subject identification numbers will be assigned sequentially within each site starting with Subject No. 1. There will be no randomization. Primary efficacy endpoint is the global response (microbiological and clinical) at the end of therapy.

Review of Inclusion/Exclusion Criteria, Medical/Disease History will be performed at Baseline. A standard 12-lead ECG will be performed at Baseline Visit or within one week prior to treatment, and at one month after the initiation of treatment. ECG will be repeated for any QTc > 450 msec for men or > 470 msec for women, or for any new cardiac signs or symptoms as clinically indicated. Apart from the ECG and pregnancy test, no other laboratory testing will be performed solely for the experimental treatment use protocol. Laboratory abnormalities which represent any clinically significant change from the baseline value (ie, a change by one toxicity grade or more) at any time during the experimental treatment use protocol period (active treatment or follow-up), which have clinical manifestations, or which require an intervention will be considered an adverse event and will be reported to the sponsor).

Baseline evaluations will be performed within 72 hours prior to the start of the investigational medication.

The investigational medication (posaconazole) will be dispensed upon completion of the Baseline assessment once there is confirmation that the Inclusion/Exclusion Criteria are met. Posaconazole is supplied as suspension 40 mg/mL (105 mL/bottle).

For seriously ill patients, posaconazole will be initially administered at a dose of 200 mg four times daily (QID) orally/enterally with meals or nutritional supplements, then once stable the regimen may be changed to 400 mg orally/enterally twice daily (BID). (Changes in dosing regimen will be at the discretion of the investigator, based on the clinical state of the patient.) Stable, ambulatory patients may be started on 400 mg PO BID. For subjects who are receiving enteral feeding, medication will be administered every six hours (QID) or every 12 hours (BID) as indicated above.

Duration of Treatment: The investigator should use discretion in determining the appropriate duration of therapy for an individual subject. Duration should be based on the following: clinical diagnosis of the invasive fungal infection; causative fungal pathogen; severity of the invasive fungal infection; severity of the subject's underlying disease; recovery from immune suppression; and rapidity of clinical response.

When the subject is discharged from the hospital, the participant will be given a supply of investigational medication (posaconazole), which will be adequate to last until the next doctor's visit. Re-supply of posaconazole will be provided at regular intervals as long as the subject completes scheduled doctor visits and continues to comply with taking posaconazole as requested, to receive maximum potential effect of the experimental medication. The experimental medication should be taken with a full meal in order to be well absorbed into the blood stream. If the medication is not well absorbed, it may be less effective.

The experimental treatment use protocol physician will examine the subject at regular scheduled clinical visits during this experimental treatment use protocol, to determine how well the subject is responding to and evaluate how well the subject is tolerating Posaconazole (SCH 56592). No extra visits are required for this experimental treatment protocol.

Specially trained pharmacists at UPMC will prepare the investigational medication. The medication will be supplied by the UPMC hospital Pharmacy and will be given to the participant by the nursing staff while the participant is in the hospital or to the care-giver, family member, spouse, an adult child, a family member or adult person responsible for caring for the subject, if discharged from hospital.

Participation in the experimental treatment protocol will continue until all signs and symptoms have resolved and ongoing therapy is no longer required to a maximum of 24 months, or until posaconazole (experimental medication) becomes commercially available (approved by the FDA). The maximum length of time a subject will be on the investigational medication will depend on type and severity of the fungal infection, response to the investigational medication and the discretion of the experimental treatment protocol doctor. For patients with complete response, posaconazole may be discontinued seven days after resolution of all signs and symptoms of infection. Subjects with Candida infections of the bloodstream, or disseminated/metastatic (deep organ) or hepatosplenic candidiasis or endocarditis should be treated with posaconazole for a minimum of 14 days or at least seven days after resolution of symptoms.

The experimental treatment use protocol will be carried out at UPMC-Presbyterian hospital. Subjects will be seen monthly and 30 days after the last dose of investigational medication to determine how well subjects are responding to the investigational medication.

ELIGIBILITY:
Inclusion Criteria:

* A proven, probable, or possible invasive fungal infection which is refractory to standard antifungal therapies after a reasonable trial of standard antifungal therapy
* A proven, probable, or possible invasive fungal infection with a prior history of serious, severe, or life-threatening toxicities related to antifungal therapy
* A proven, probable, or possible invasive fungal infection with documented organ dysfunction (such as renal dysfunction defined as serum creatinine > 2.5 mg/dL or estimated creatinine clearance < 25 mL/minute), which precludes the continued administration of standard antifungal therapy
* A proven or probable invasive fungal infection for which there are currently no other clinically reasonable effective therapies
* A history of a proven or probable invasive fungal infection previously treated with posaconazole in a chronically immunosuppressed patient that requires oral antifungal suppressive therapy.
* A proven or probable invasive fungal infection in patients who have failed a reasonable trial of other licensed antifungal agents, either due to progression or lack of improvement of the infection
* A history of proven or probable invasive fungal infection in patients requiring ongoing antifungal therapy as chronic maintenance after initial control of disease with other antifungal agents, but who have become intolerant to licensed azoles. In these cases where long term parenteral antifungal therapy (e.g., amphotericin B or echinocandins) is not considered practical or clinically reasonable by the physician, posaconazole may be considered to be a potential treatment option.
* Patients with debilitating but no immediately life threatening fungal diseases, where significant morbidity may result in disability and where prior antifungal therapy has been unsuccessful (e.g., chronic candidiasis with dehydration and malnutrition, or cutaneous phaeohyphomycosis and mycetoma).

Exclusion Criteria:

* Females who are pregnant or who continue to breast feed infants.
* History of serious or severe hypersensitivity or idiosyncratic reactions to azole antifungals
* Subjects who require ongoing treatment with any prohibited medication and for whom an appropriate washout period has not elapsed. Those drugs known to interact with azoles and that may lead to life-threatening side effects: terfenadine, cisapride, and ebastine at entry or within 24 hours before entry, or astemizole at entry or within 10 days before entry; those known to lower the serum concentration/efficacy of azole antifungal agents: cimetidine, rifampin, carbamazepine, phenytoin, rifabutin, barbiturates, and isoniazid at entry or within 24 hours before entry; and those receiving vinca alkaloids, or anthracyclines with evidence of cardiotoxicity.
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the experimental treatment use protocol, ie, any condition requiring the use of prohibited drugs or unstable medical conditions other than a hematological disorder such as unstable cardiac disorder (including acute myocardial infarction or unstable myocardial ischemia/angina within 30 days, ventricular arrhythmia within 30 days, uncontrolled atrial fibrillation, or atrial fibrillation/flutter with symptomatic bradycardia [sick sinus syndrome], or unstable congestive heart failure) or impairment expected to be unstable or progressive during the course of this experimental treatment use protocol (eg, recurrent or uncontrolled seizure disorders, demyelinating syndromes, or progressive peripheral neuropathy).
* Subjects receiving vinca alkaloids or anthracyclines within 24 hours of enrollment or requiring therapy with vinca alkaloids or anthracyclines within the next 30 days for treatment of uncontrolled (pre-existing) malignancy or requiring ongoing therapy with vinca alkaloids or anthracyclines
* Subjects requiring ongoing systemic antifungal agents in addition to investigational medication (combination use is not permitted without prior authorization of the sponsor project physician).
* Subjects with an ECG with QTc interval greater than 450 msec for men, and greater than 470 msec for women at entry or within seven days prior to entry
* Any condition requiring the use of prohibited drugs
* Hepatic function tests: alanine amino transferase (ALT) or aspartate amino transferase (AST) > 10 times upper limit of normal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2004-08; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
provide posaconazole to patients with invasive fungal infections

SECONDARY OUTCOMES:
posaconazole where no other drug is commercially available

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Hardalo, MD, Principal Investigator — Schering-Plough
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States